CLINICAL TRIAL: NCT06859853
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MWN109 Injection in Healthy Subjects
Brief Title: A Study to Evaluate MWN109 Injection in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Minwei Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MWN109-101
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Overweight or Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Drug: Subcutaneous single and mutiple dose
- MWN109 injection (Active Comparator): * Participants in SAD cohorts will be randomized to receive MWN109 injection or placebo across 5 cohorts. Planned dosage per cohorts are A1:0.25mg, A2:0.75mg, A3:1.5mg, A4:3.0mg, A5:6.0mg.
  * Participants in MAD cohorts will be randomized to receive MWN109 injection or placebo across 4 cohorts. The IP will be administered via SC injection once weekly (QW) for approximately 4 doses. Planned dosage per cohorts are: B1-1.5 mg/1.5 mg/1.5 mg/1.5 mg; B2-1.5 mg/3.0 mg/3.0 mg/3.0 mg; B3-1.5 mg/3.0 mg/4.5 mg/6.0 mg; B4-1.5 mg/3.0 mg/6.0 mg/9.0 mg.
  Interventions: Drug: Placebo; Drug: Subcutaneous single and mutiple dose

INTERVENTIONS:
Drug: Placebo — Sub cutaneous injection on the abdomen by a qualified member of study staff.
Drug: Subcutaneous single and mutiple dose — Sub cutaneous injection on the abdomen by a qualified member of study staff.

SUMMARY:
This study is a Phase1, randomized, double-blinded, and placebo-controlled study. In each cohort, enrolled participants will be randomized to receive either placebo or MWN109.

DETAILED DESCRIPTION:
A total of 72 healthy volunteers are expected to be enrolled into this study. Study consists of 2 parts- Part A- Single Ascending dose (SAD) and part B- Multiple ascending dose (MAD).

The entire study duration per participant is estimated to be a maximum of 8 weeks for the single ascending dose (SAD) part and 12 weeks for the multiple ascending dose (MAD) part. The end of study is defined as the date of the last visit of the last participant in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, aged 18 to 50 years (inclusive) at Screening.
2. [Part A: SAD] BMI of 19.0 to 40.0 kg/m2 (inclusive). [Part B: MAD] BMI of 27.0 to 45.0 kg/m2 (inclusive) with a minimum body weight of 50.0 kg for females and 55.0 kg for males.
3. History of stable body weight for 3 months (defined as change < 5%).
4. Resting heart rate (supine) ≥ 45 bpm and ≤ 90 bpm with a single 12-lead ECG at Screening.
5. Females of childbearing potential and males will agree to use contraception as detailed further in the protocol.
6. Male participants must agree to refrain from sperm donation and females should refrain from ova donation from D-1 until 4 months after the last administration.
7. Able to comprehend and willing to sign an ICF and to abide by all study requirements and restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any cardiovascular, metabolic, allergic, endocrine, renal, hepatic, gastrointestinal, hematological, pulmonary, respiratory, dermatological, neurological, gynecological, psychiatric, disorders as determined by the investigator (or designee).
2. History of pheochromocytoma or has uncontrolled blood pressure, as defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg.
3. History of insulinoma or has an event of blood glucose < 2.8 mmol/L within 1 year prior to Screening, or with ≥ 3 times of hypoglycemia symptoms within 3 months prior to Screening.
4. History of febrile illness within 7 days prior to the first dose of IP or participants with evidence of active infection.
5. Any of the following:

   1. QTcF > 450 msec regardless of gender , confirmed by repeat measurement.
   2. QRS duration > 110 msec confirmed by repeat measurement.
   3. PR interval > 220 msec confirmed by repeat measurement.
   4. Findings which would make QTc measurements difficult or QTc data uninterpretable.
   5. History of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome).
6. Known history or family history of thyroid C-cell tumor/carcinoma, multiple endocrine neoplasia syndrome type 2 (MEN2), thyroid dysfunction or thyroid hormone abnormality.
7. History of diabetes mellitus Type I or II or clinical evidence of diabetes (e.g., hemoglobin A1c ≥ 6.5%, fasting blood glucose ≥ 126 mg/dL [7.0 mmol/L]) at Screening, non-fasting glucose ≥ 200 mg/dL (11.1 mmol/L) at Screening, or use of any hypoglycemic drugs during Screening or within 3 months prior to Screening
8. History of acute or chronic pancreatitis, symptomatic gallbladder disease, pancreatic injury and other high-risk factors that may lead to pancreatitis.
9. With any of following laboratory abnormality:

   1. Elevation in serum amylase or lipase (> 1.5 × upper limit of normal [ULN]).
   2. Have serum AST or ALT > 2 × ULN or total bilirubin >1.5 × ULN.
   3. Have serum TG ≥ 5.65 mmol/L (500 mg/dL) at screening
   4. Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m2.
10. History of clinically significant abnormal gastric emptying (e.g., gastric outlet obstruction, gastroparesis), severe chronic gastrointestinal diseases (e.g., having active ulcer within 6 months prior to Screening, active gastritis or esophagitis, or uncontrolled gastroesophageal reflux disease, irritable bowel disease or severe inflammatory bowel disease).
11. Long-term use of drugs directly affecting the gastrointestinal motility (including but not limited to mosapride, cisapride) or gastrointestinal surgery within 12 weeks prior to Screening and are inappropriate for participation in this clinical study as assessed by the Investigator.
12. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), or human immunodeficiency virus (HIV-1 and HIV-2) antibodies and p24 antigen.
13. Any history of severe psychiatric disorder such as major depressive disorder, bipolar disorder, and schizophrenia, or history of suicidal ideation, behavior or attempts or other psychiatric disorder (within 2 years of Screening).
14. Any suicidal ideation as identified by endorsement of (answered yes to) any of the items numbered 1-5 on the Columbia Suicide Severity Rating Scale (C-SSRS), if applicable.
15. History of alcoholism or drug/chemical abuse within 1 year prior to D-1.
16. Alcohol consumption of > 21 units per week for males and > 14 units per week for females, on average. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
17. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) during the Screening period.
18. Daily use of more than 10 cigarettes/day (on average), or 2 cigars/day (on average), or equivalent use of any tobacco product within 6 weeks prior to Screening.
19. Females of pregnant or lactating, or those with a positive pregnancy test at Screening.
20. Intolerance to venipuncture for blood sampling or history of fainting at blood drawing or sight of blood, unless deemed acceptable by the Investigator (or designee).
21. History of severe Types I-IV hypersensitivity reactions, anaphylaxis, cytokine release syndrome, atopic individuals, or allergic reactions to multiple drugs. If the Investigator is considering enrolling a participant with drug allergies, agreement with the Medical Monitor should be sought.
22. History of or suspected allergy or hypersensitivity to the investigational product or its components
23. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
24. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to D-1, unless deemed acceptable by the Investigator (or designee).
25. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to D-1, unless deemed acceptable by the Investigator (or designee).
26. Participants with a history of infectious diseases (which may affect the ability of the participant to participate in the study at the discretion of the Investigator), severe trauma, or major surgical operation within 4 weeks prior to Screening.
27. Have been vaccinated within 4 weeks prior to Screening or plan to have vaccination during the study.
28. Donation of blood or massive blood loss (> 450 mL) OR receipt of blood products within 12 weeks prior to Screening.
29. Participation in a clinical study involving administration of an investigational agent/device or vaccine (new chemical entity) or having received a biological product within 12 weeks prior to Screening.
30. Poor peripheral venous access.
31. Are investigative site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
32. The presence of clinically significant physical examination, vital sign, drug, or ECG findings at Screening or baseline or laboratory findings at Screening that, in the opinion of the Investigator or Medical Monitor, may interfere with any aspect of study conduct or interpretation of results.
33. Any skin condition and/or tattoo that may interfere with the evaluation of safety at the injection site.
34. Are deemed unsuitable by the Investigator (or designee) for any other reason.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Incidence of treatment emergent adverse events (TEAEs) following treatment administration | Part A- Up to Day 29; Part B- Up to Day 50 post first dose administration
Number of participants with change in laboratory parameters following treatment administration | Part A- Up to Day 29; Part B- Up to Day 50 post first dose administration
  Changes in clinical laboratory parameters include urine drug screening, alcohol breath test. serum virology, pregnancy test. hematology, blood chemistry, urinalysis, coagulation function, and thyroid function.
Number of participants with change in Vital signs following treatment administration | Part A- Up to Day 29; Part B- Up to Day 50 post first dose administration
  Vital signs include measurement of heart rate (HR) respiration rate (RR), systolic and diastolic blood pressure (BP) and body temperature.
Incidence of anti-drug antibody (ADA) formation following treatment administration | Part A- Up to Day 29; Part B- Up to Day 50 post first dose administration

SECONDARY OUTCOMES:
PK parameters- Cmax: maximum observed concentration | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- -Tmax: time to reach maximum concentration | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- t½: half-life | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- AUC0-inf: area under the concentration-time curve from time zero to the theoretical infinite time | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- AUCo-t: area under the concentration-time curve from time zero to the time of the last quantifiable concentration | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- AUC0-168h: area under the concentration-time curve from time zero to 168 h post dose | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- CL/F: apparent clearance | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- Vd/F: apparent volume of distribution | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.
PK parameters- MRT: mean residence time | SAD- Up to Day 29; MAD- Up to Day 50 post first dose administration.

CONTACTS AND LOCATIONS:
Overall Officials: Guitao Zhang, Study Chair — Shanghai Minwei Biotechnology
Locations (1):
- Veritus Research, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No